CLINICAL TRIAL: NCT02264418
Title: Safety and Tolerability of Single and Repeated Doses of ODM-203: An Open-label, Non-randomised, Uncontrolled, Dose Escalation, Multicentre, First-in-Human Study in Subjects With Advanced Solid Tumours
Brief Title: Safety and Tolerability of ODM-203 in Subjects With Advanced Solid Tumours
Acronym: KIDES-203
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3113001
Record Dates: First submitted 2014-09-19; First posted 2014-10-15 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumours
Keywords: Solid tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ODM 203 (Experimental): Oral capsules given once daily dosage 50-800mg
  Interventions: Drug: ODM 203
- ODM-203 (Experimental): Oral tablets given once daily 200-1600mg
  Interventions: Drug: ODM 203

INTERVENTIONS:
Drug: ODM 203 — ODM 203
  Arms: ODM 203
Drug: ODM 203 — ODM 203

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety and tolerability of escalating doses of ODM-203 in subjects with advanced solid tumours and to determine the maximum tolerated dose and dose limiting toxicities.

DETAILED DESCRIPTION:
The safety profile of ODM-203 will be explored together with the pharmacokinetics, pharmacodynamics and tumour response to treatment with ODM-203 to recommend the dosing regimen for further clinical studies. The pharmacokinetic properties of ODM 203 will be evaluated after single and multiple dose administrations at different dose levels

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female subjects over 18 years of age
* Subjects with histologically or cytologically confirmed locally advanced or metastatic tumours. Subjects in Part 2 to have a tumour/genetic aberration.
* Availability of tumour sample for genetic analysis
* Adequate haemopoietic, hepatic and renal function
* Eastern Cooperative Oncology Group performance status of 0 to 1
* Serum mineral levels phosphate: 2.5 mg/dl; calcium: 8.8 mg/dl; magnesium: 1.2 mg/dl; potassium: 11.7 mg/dl; sodium: 299mg/dl.
* Recovery from reversible adverse events of previous systemic anti-cancer therapies to baseline or grade 1 with the exception of alopecia;stable neuropathy of grade 2 induced by previous cancer treatment
* Life expectancy of 12 weeks or more

Exclusion Criteria:

* Any prior anti VEGFR/FGFR treatment related AE that in the judgement of the investigator is considered severe/life threatening
* Subjects receiving warfarin
* Active central nervous system metastases not controlled by prior surgery/radiotherapy and/or low dose steroids for 4 weeks or more
* Subjects with current evidence of endocrine alteration of calcium-phosphate homeostasis
* Concomitant therapies known to increase serum phosphorus and/or calcium levels that cannot be discontinued or switched to a different therapy are not permitted within 14 days before the first dose of ODM-203.
* Significant cardiovascular conditions/circumstances as follows:
* a active or unstable cardio/cerebro-vascular disease
* b Uncontrolled hypertension (systolic blood pressure ≥ 150mmHg and/or diastolic blood pressure ≥ 90mg Hg with optimised antihypertensive therapy.
* c history of severe arrhythmia, familial arrhythmia, conduction abnormality or congenital long QT syndrome
* dConcomitant therapies known to prolong the QT interval and associated with a risk of Torsades de Pointes are not permitted within 7 days before the first dose of ODM 203
* e Repeatable prolongation of QTcF interval ≥ 450 msec or any clinically significant abnormality in the ECG at screening in 2 out of 3 recordings
* f Left ventricular ejection fraction <50% at screening
* Subjects who received systemic anticancer treatment prior to the first dose of ODM-203 within the following timeframes: less than 28 days since the last dose of antineoplastic therapy and/or 28 days of wide field radiotherapy or 14 days of limited field radiation for palliation
* Major surgery or serious infection within 21 days of the first dose of ODM-203
* Known gastrointestinal disease or a procedure that may affect absorption of ODM 203
* Serious concurrent medical condition or psychiatric illness
* History and/or current evidence of ectopic mineralisation/calcification
* Known active or past history of other primary malignancy
* Female of child bearing potential
* Female of child bearing potential or male subject with a female partner of child bearing potential who does not agree to use effective contraception during the study and for 3 months after the last dose of ODM 203
* Known hypersensitivity to the study treatment excipients
* Any condition which in the opinion of the investigator would impair the subject's ability to comply with the study procedures
* Participation in another interventional clinical trial/ concurrent treatment with any investigational drug within 4 weeks prior to the start of treatment with ODM 203

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | From the date of informed consent to the date of the end of study visit estimated to be 6 months
  Number of adverse event counts

SECONDARY OUTCOMES:
Frequency of responders to Response evaluation criteria in solid tumours (RECIST) | Subjects will be followed for the duration of time in the study, expected to be an average of 6 months
  The frequency of responders according to RECIST will be evaluated by dose level.
Eastern Cooperative Oncology Group (ECOG) Performance status | Subjects will be followed for the duration of time in the study, expected to be an average of 6 months
  The ECOG performance status and the change from baseline will be reported by dose level.
Area under the plasma concentration curve (AUC) | 0 to 24hours post dose Day 1 and Day 15
  Area under the plasma concentration curve (AUC) of ODM-203 will be measured to evaluate the relationship between ODM-203 dose, plasma exposure, pharmacodynamics and safety
Peak plasma concentration (Cmax) | After first dose administration to 24 hours Day 1 and Day 15
  Peak plasma concentration (Cmax) of ODM-203 will be measured to evaluate the relationship between ODM-203 dose, plasma exposure, pharmacodynamics and safety

CONTACTS AND LOCATIONS:
Overall Officials: Petri Bono, MD, Principal Investigator — Helsinki University Central Hospital
Locations (8):
- Finsen Centre, Copenhagen, Denmark
- Helsinki University Central Hospital, Department of Oncology, Helsinki, Finland
- France (2):
  - Institut Bergonie, Bordeaux
  - Gustave Roussy Oncology Institute, Villejuif
- European Institute of Oncology, Milan, Italy
- Vall d'Hebron University Hospital, Barcelona, Spain
- United Kingdom (2):
  - Sarah cannon Research Institute, London
  - UCL Cancer Institute, London

REFERENCES:
- [Derived] Bono P, Massard C, Peltola KJ, Azaro A, Italiano A, Kristeleit RS, Curigliano G, Lassen U, Arkenau HT, Hakulinen P, Garratt C, Ikonen T, Mustonen MVJ, Rodon JA. Phase I/IIa, open-label, multicentre study to evaluate the optimal dosing and safety of ODM-203 in patients with advanced or metastatic solid tumours. ESMO Open. 2020 Dec;5(6):e001081. doi: 10.1136/esmoopen-2020-001081. PMID 33262202